CLINICAL TRIAL: NCT02238912
Title: Evaluation of Preclinical Toxicity of a Siddha Formulation Kandhaga Rasayanam ( KR ) and Its Therapeutic Efficacy in Padarthamarai ( Dermatophytoses ) by an Open Clinical Trial
Brief Title: Evaluation of Preclinical Toxicity andTherapeutic Efficacy of Kandhaga Rasayanam in Padarthamarai
Acronym: KR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National institute of Siddha (Other Government)
Responsible Party: Principal Investigator, Dr.R.Meena, PhD Research scholar, National institute of Siddha
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXII(1)/29097/2011
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Tinea Infections Such as Tinea Corporis, Tinea Cruris, Tinea Pedis, Tinea Mannum, Tinea Barbae, Tinea Capitis Are Studied
Keywords: tinea
MeSH Terms: conditions — Tinea Cruris; Tinea Pedis; tinea barbae; Tinea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kandhaga Rasayanam- single arm (Experimental): Kandhaga Rasayanam- 2grams twice a day for 45 days
  Interventions: Drug: kandhaga rasayanam

INTERVENTIONS:
Drug: kandhaga rasayanam — KANDHAGA RASAYANAM is a siddha herbo mineral drug with sulphur as a sole mineral ingredient. It is chosen from the classic Siddha text Siddha Vaidhya Thirattu.
  Other Names: Siddha herbo mineral drug KR.

SUMMARY:
this study is intended to find out the therapeutic efficacy of the siddha drug Kandhaga Rasayanam in Padarthamarai ( Ring worm infection )

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed with tinea infection.
* direct microscopy skin scraping test positive.

Exclusion Criteria:

* pregnant or nursing women.
* use of other topical or oral antifungals, immunosuppressive drugs, anthelmintic drugs either currently or during 2 weeks preceeding initiation of drug trial.
* allergy or hyperensitivity to any component of the drug.
* clinical case of eczema, lichen planus, pityriasis versicolor, drug induced eruptions, urticaria, intertrigo, tinea ungium.
* diabetic patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
skin scrapping test | 45 days

SECONDARY OUTCOMES:
itching, quality of life | 45 days

OTHER OUTCOMES:
burning sensation, vanishing of lesions | 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- National institute of siddha, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] AYUSH PORTAL, GOOGLE SCHOLAR
- See also: TRIAL REGISTERED IN CTRI — http://www.ctri.nic.in/